CLINICAL TRIAL: NCT00431093
Title: A Multicenter, Randomized, Double-Blind, Double Dummy, Group-Comparative Trial to Compare the Effects of Livial® and Activelle ® on the Vaginal Bleeding Pattern, Vasomotor Complaints, Vaginal Atrophy, QoL and Sexual Function
Brief Title: Trial to Compare the Effects of Tibolone (Livial®) and Continuous Combined Low-Dose Estradiol/Noresterone (Activelle®)
Acronym: TOTAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P06673; C-1755 (Other: Schering-Plough)
Record Dates: First submitted 2007-02-02; First posted 2007-02-05 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Menopause
MeSH Terms: interventions — tibolone; Estradiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): tibolone
  Interventions: Drug: low-dose estradiol/noresterone
- 2 (Active Comparator): low-dose estradiol/noresterone
  Interventions: Drug: tibolone

INTERVENTIONS:
Drug: tibolone — uncoded tablets, at a dose of 2.5 mg per tablet; Subjects were to take 1 Livialâ tablet and 1 -matched Activelleâ placebo tablet, orally, once a day (preferably at the same time).
  Other Names: Livial
  Arms: 2
Drug: low-dose estradiol/noresterone — Activelleâ, estradiol (E2) 1 mg and norethisterone acetate (NETA) 0.5 mg per tablet, was supplied as uncoded tablets.
  Subjects were to take 1 Activelleâ tablet and 1 Livialâ-matched placebo tablet, orally, once a day (preferably at the same time).
  Other Names: Activelle®
  Arms: 1

SUMMARY:
The present trial is undertaken to compare the effects of Tibolone with a low-dose HRT regimen.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be healthy and postmenopausal women, >= 45 and < 65 years of age, with an intact uterus.
* Subjects must have been postmenopausal for less than 15 years.
* Body Mass Index >18 and =< 32 kg/m2.
* Voluntary written informed consent is required.

Exclusion Criteria:

* Any unexplained abnormal uterine bleeding after the menopause.
* Double layer endometrial thickness = 6 mm as assessed by transvaginal ultrasonography.
* Treatment with oral estrogen and/or progestogen therapy within 4 weeks prior to screening, or treatment with transdermal therapy and local estrogen applications within 4 weeks prior to screening.
* Any previous or current unopposed estrogen administration, prior use of estrogen pellets or tamoxifen citrate (occasional use of estrogen-containing vaginal cream is allowed after the appropriate wash-out period is completed). Estrogen combined with sequential administration of progestogen should have been at least 10 days per 28 day cycle.
* The following wash-out periods apply:

  * 4 weeks for transdermal hormonal treatment, local estrogen applications or other non-hormonal medication known to act on the relief of vasomotor symptoms (e.g. clonidine)
  * 4 weeks for phytoestrogens, tibolone, intra-uterine or oral progestogen and oral estrogen/progestogen therapy
  * 6 months for progestogen implants or injections and estrogen/progestogen injectable therapy.
* Any subjects who are either using phytoestrogens, tibolone, intra-uterine or oral progestogen, progestogen implants or injections, estrogen/progestogen combination therapy or any other non-hormonal medication known to act on the relief of vasomotor symptoms and who have not observed the appropriate wash-out periods (see previous exclusion criteria).
* Any serious disease or disorder; or any endocrine disorder; (controlled hypo/hyperthyroidism and diabetes mellitus Type II is allowed).
* Diseases for which exogenous hormonal steroids are contraindicated.
* History or presence of any malignancy, except successfully treated nonmelanoma skin cancers.
* History or presence of cardiovascular or cerebrovascular conditions:

  * thrombophlebitis, thrombosis or thromboembolic disorders.
* History or presence of liver, gallbladder (subjects who have had a cholecystectomy will not be excluded) or renal disease, epilepsy or classical migraine headaches.
* History or presence of clinically significant depression or other psychiatric disorders which, in the investigator's judgment, might compromise or confound the subject's participation in the trial.
* Uncontrolled high blood pressure: systolic pressure > 170 mmHg and/or diastolic pressure > 105 mmHg, measured after 5 minutes in a sitting position.
* Abnormal cervical Pap smear (corresponding to PAP = III, or LSIL, HSIL, ASCUS, AGCUS in the Bethesda classification)
* Abnormal, clinically significant results of the mammography.
* Presence of fibrocystic disease of the breast.
* Presence of otosclerosis.
* Known hypersensitivity to any of the ingredients of the trial medication.
* Any subjects using either steroids, drugs known to affect sexual functioning and mood (antidepressants, psychoactive drugs, sedatives, neuroleptics, narcotics, benzodiazepines), drugs know to interfere with the pharmacokinetics of the steroids (hydantoins, primidone, rifampicin, barbiturates, carbamazepine, griseofulvin, warfarin, ketoconazole, or products containing St. John's wort), or raloxifene hydrochloride. A wash-out period of 4 weeks will apply to subjects using these drugs. Sporadical use of benzodiazepines (twice or less a week) is allowed

Ages: 45 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 570 (Actual)
Dates: Start 2002-11; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
For the bleeding evaluation, subject will be given a diary card to record the days on which no bleeding, vaginal spotting or bleeding occurs | starting from baseline and during the whole trial period.

SECONDARY OUTCOMES:
Hot flushes recorded on a daily diary card during the whole trial period. | Entire trial
A mammography to assess breast density and blood samples to determine the changes in endocrine parameters. | screening and week 48
A vaginal smear to assess the Vaginal Maturation Index and the Karyopycnotic Index results | Baseline and week 48
Urogenital complaints assessed with the Local Urogenital Complaints Rating Scale. | At baseline, week 12, week 24 and week 48
Health-related quality of life measured with the Women's Health Questionnaire 36-items (WHQ-36) the McCoy Female Sexuality Questionnaire-Short Form 9-items (MFSQ-SF) collecting prospectively medical resources utilization items | At baseline and week 48

REFERENCES:
- [Derived] Hammar ML, van de Weijer P, Franke HR, Pornel B, von Mauw EM, Nijland EA; TOTAL Study Investigators Group. Tibolone and low-dose continuous combined hormone treatment: vaginal bleeding pattern, efficacy and tolerability. BJOG. 2007 Dec;114(12):1522-9. doi: 10.1111/j.1471-0528.2007.01537.x. PMID 17995496